CLINICAL TRIAL: NCT04609722
Title: Effect of Solution-Focused Support Program on Anxiety Levels of Parents With Children Aged 3-6 Years During the COVID-19 Pandemic
Brief Title: Effect of Solution-Focused Support Program on Anxiety Levels of Parents During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Mürşide Zengin, Adıyaman University, Adiyaman University Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020/751
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Anxiety; Parents; Covid19
Keywords: anxiety; child; nursing practice; parents; Solution-Focused Support Program
MeSH Terms: conditions — Anxiety Disorders; COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Solution-Focused Support Program will apply to the participants.
  Interventions: Other: Solution-Focused Support Program
- control group (No Intervention): No intervention will be applied to the parents in the control group.

INTERVENTIONS:
Other: Solution-Focused Support Program — All participants will be given a program of 4 sessions for 4 weeks. Each session is planned to last approximately 50 minutes.
  Arms: intervention group

SUMMARY:
In this research, it was aimed to determine the anxiety levels of parents in the Covid-19 pandemic and to examine the effects of the Solution-Focused Support Program, which is planned to be given to parents with high anxiety levels.

DETAILED DESCRIPTION:
The study is conducted with parents whose children aged 3-6 years, and have high anxiety levels. In collecting research data; an introductory information form prepared by researchers and the State-Trait Anxiety Inventory will be used.

ELIGIBILITY:
Inclusion Criteria:

* Parents with children aged 3-6,
* Having internet at home or mobile phone,
* Parents who volunteer to participate in the study

Exclusion Criteria:

* Having communication problems,
* Parents who have not attended at least one session

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | 5 minutes
  STAI was developed by Spielberg et al. In 1970 to measure the trait and state anxiety levels of individuals and was adapted to Turkish by Öner and Le Compte (1983) (Gilik and Avşaroğlu 2017). There are a total of 40 questions in the State-Trait Anxiety Scale. The State Anxiety Sub-Scale (STAI-S) evaluates how an individual feels at a particular time and under certain conditions. The Trait Anxiety Subscale (STAI-T) generally assesses how an individual feels. The scores obtained from both scales vary between 20 and 80. High score indicates high anxiety level, low score indicates low anxiety level.

CONTACTS AND LOCATIONS:
Overall Officials: Ceyda Başoğul, Principal Investigator — Adiyaman University; Emriye Hilal Yayan, Principal Investigator — İnönü University; Mürşide Zengin, Principal Investigator — Adiyaman University
Locations (1):
- Online- Data will be collected through the form created with the Google-Forms, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No